CLINICAL TRIAL: NCT06248788
Title: Study to Survey the Normal Range of Salivary Immunoglobulin A (sIgA) Levels Measured by a Point of Care Device in Healthy Adult Women and Men
Brief Title: Salivary Immunoglobulin A (sIgA) Normal Range Study
Acronym: sIgA
Status: Completed | Type: Observational
Sponsor: 4Life Research, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: RSC-014-00
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Salivary Immunity
Keywords: salivary immunoglobulin A; point of care device

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: PoC Device — PoC Device for Testing Salivary IgA

SUMMARY:
Salivary Immunoglobulin A (sIgA) is a marker of immune system activity. Typically, sIgA is determined by an ELISA test in which samples have to be sent to a specialized laboratory for testing. Investigators have developed a new instrument that is small, portable, and easy to use. This instrument is available for consumers to purchase and test their own sIgA at home.

ELIGIBILITY:
Inclusion Criteria:

* Adults committed to attend the session and follow the instructions described in Experimental Design will be included.

Exclusion Criteria:

* Participant with mouth infection or oral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: any adults that are free from oral infections or oral diseases
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Salivary IgA | 0 minute

CONTACTS AND LOCATIONS:
Locations (1):
- 4Life Research, Sandy City, Utah, United States

IPD SHARING:
Plan to Share IPD: No